CLINICAL TRIAL: NCT06888999
Title: In Vitro Exposure by VR to Enhance Return to Work After Sick Leave Due to Mental Health Related Complaints
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: KLM Royal Dutch Airlines (Unknown); KLM Health Services (Unknown); Villa Uitzicht (Unknown)
Responsible Party: Principal Investigator, Roosmarijn Schelvis, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025.0183
Record Dates: First submitted 2025-03-20; First posted 2025-03-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Return to Work; Occupational Stress; Self-Efficacy
Keywords: virtual reality; return to work; pilot randomized controlled trial; cabin crew; stress; return to work self-efficacy; job anxiety; usability; return to work attitude
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing an intervention group with a care as usual group. Randomization is carried out at the individual level.
Masking Description: Due to the intervention, it is not possible to blind researchers, case provides, investigators and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual plus VR (Experimental): Participants in the intervention group receive care as usual from the occupational physician and a psychologist and participate (al least once) in a VR-session. During the VR-session, guided by the psychologist, participants are virtually exposed to their workplace.
  Interventions: Other: In vitro exposure to workplace by VR plus care as usual
- Care as usual (Active Comparator): Participants in the care as usual group receive care as usual from the occupational physician and a psychologist.
  Interventions: Other: Care as usual: Guidance from occupational physician and psychologist focused on returning to work

INTERVENTIONS:
Other: In vitro exposure to workplace by VR plus care as usual — During the VR-session, guided by the psychologist, participants are virtually exposed to their workplace using VR glasses. Based on the experience of the participants during the vitual visit to their workplace, the psychologist can adjust the therapy. In addition care as usual is provided (see description active comparator).
  Arms: Care as usual plus VR
Other: Care as usual: Guidance from occupational physician and psychologist focused on returning to work — Guidance by the occupational physician and a psychologist from a psychologist practice specialized in counseling cabin crew and guiding them with returning to work.
  Arms: Care as usual

SUMMARY:
The goal of this pilot randomised controlled trial is to investigate whether in vitro exposure by VR enhances return to work (RTW) in flight cabin crew on sick leave with mental health related complaints. The main research questions are: 1. Does VR enhances time to RTW? 2. Does VR increase self-efficacy and positive cognitions regarding RTW, and decrease job anxiety? Researchers will compare a control group receiving care as usual as provided by the occupational physician and a psychologist to an intervention group receiving care as usual plus (al least) one session with VR-glasses in which participants are virtually exposed to their workplace.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of in vitro exposure to the workplace by means of VR to decrease time to RTW of sick-listed flight cabin crew with mental health related complaints compared to usual care. The study design is a pilot randomized controlled trial, including an intervention and control group. Sick-listed workers in the control group receive care as usual from the occupational physician and a psychologist. Sick-listed workers in the intervention group receive care as usual from the occupational physician and a psychologist and participate in a VR-session. During the VR-session, guided by the psychologist, participants are virtually exposed to their workplace. Data on the primary outcome of RTW is collected based on the register data from the occupational health service (6 and 12 months after baseline). Data on secondary outcomes (self-efficacy, cognitions regarding RTW and job anxiety) is collected with baseline and follow-up questionnaires (4 months after baseline).

ELIGIBILITY:
Inclusion Criteria:

- sick listed cabin crew with mental health related complaints that are referred by the occupational physician to a specific psychotherapist practice

Exclusion Criteria:

* epilepsy
* vestibular disorder
* no signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Time to RTW | 6 months and 12 months after baseline
  Time between start of sickness absence until participant is considered 'fit to fly' by the occupational physician, measured by register data from the occupational health service.

SECONDARY OUTCOMES:
Stress-related complaints | Baseline and 4-months follow-up
  Stress-related complaints (e.g., type of disease, severity of symptoms) by means of Perceived Stress Scale (PSS-10). The PSS-10 consists of 10 items rated on a 5-point Likert scale, ranging from 0 (never) to 4 (very often). A high score means more stress-related complaints
Self-efficacy regarding return to work | Baseline and 4-months follow-up
  Self-efficacy regarding return to work measured by Return-to-Work Self-Efficacy scale (RTW-SE). The RTW-SE contains of 11 items. The items are rated on a five point scale The response categories vary from 1 (totally disagree) to 6 (totally agree). A high score means more return to work self-efficacy
Attitude regarding return to work | Baseline and 4-months follow-up
  Scale on attitude regarding return to work. Attitude regarding return to work is measured with a 8-item scale measuring the attitude towards working again. The items are rated on a 4-point scale ranging from 1 (disagree very strongly) to 4 (agree very strongly). A higher score means a more positive attitude towards return to work.
Job anxiety | Baseline and 4-months follow-up
  Anxiety related to the job measured by the Job Anxiety Scale. The items are rated on a 5-point Likert scale, ranging from of 0 (no agreement) to 4 (full agreement). A higher score means more job anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Roosmarijn M.C. Schelvis, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- KLM Health Services, Schiphol, Netherlands

IPD SHARING:
Plan to Share IPD: No
We will not publish the complete dataset to protect the privacy of the participants.

REFERENCES:
- [Background] Schmalbach I, Schmalbach B, Kalkbrenner A, Bassler M, Hinz A, Petrowski K. Psychometric properties of the job anxiety scale. Front Psychol. 2023 Apr 25;14:1020596. doi: 10.3389/fpsyg.2023.1020596. eCollection 2023. PMID 37179888
- [Background] Muschalla B, Linden M, Olbrich D. The relationship between job-anxiety and trait-anxiety--a differential diagnostic investigation with the Job-Anxiety-Scale and the State-Trait-Anxiety-Inventory. J Anxiety Disord. 2010 Apr;24(3):366-71. doi: 10.1016/j.janxdis.2010.02.001. Epub 2010 Feb 11. PMID 20207103
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417